CLINICAL TRIAL: NCT07220148
Title: Multimodal Assessment of Neural, Neuroendocrine, and Immune Cue Responses in Binge Drinkers in the Laboratory and Real World
Brief Title: Multimodal Immune and Neuroendocrine Assessment in Drinkers
Acronym: MIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Sara K Blaine, Associate Professor, Auburn University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000843
Record Dates: First submitted 2025-10-19; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; Laboratories

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binge Drinkers (Experimental): Behavioral Intervention: Laboratory alcohol administration and cue exposure task; completion of EMA and blood sampling at all waves.
  Interventions: Behavioral: Alcohol Cue Reactivity and Laboratory Alcohol Administration Paradigm
- Social Drinkers (Experimental): Behavioral Intervention: Identical procedures without the binge-level drinking phenotype; completion of EMA and blood sampling at all waves.
  Interventions: Behavioral: Alcohol Cue Reactivity and Laboratory Alcohol Administration Paradigm

INTERVENTIONS:
Behavioral: Alcohol Cue Reactivity and Laboratory Alcohol Administration Paradigm — Mechanistic evaluation of neural, neuroendocrine, and immune biomarkers underlying alcohol cue reactivity and drinking behavior.

SUMMARY:
The goal of this clinical trial is to better understand how blood flow in the brain, levels of the hormone, cortisol, and levels of an immune factor, interleukin-6, change in response to pictures of alcohol versus water pictures of water in healthy people who regularly consume alcohol. Researchers will learn about how the brain processes our environment and how it relates to people's drinking behaviors. This information is important because it may allow us to develop new treatments for Alcohol Use Disorders.

Participants will be asked to fill out psychological questionnaires at the first appointment. Then, they will do MRI scans with blood draws at visits 2-6. After each MRI scan, participants will undergo the Alcohol Taste Test, which involves drinking beer.

There will be a total of 3 visits at baseline, 2 visits one year later, and 2 visits one year after that. Each visit will last 2 hours. Each year, participants will do 21 days of surveys on a smart phone (4 surveys a day; each survey takes less than 2 minutes). The total time commitment for the entire study will be 23 hours.

ELIGIBILITY:
Inclusion Criteria:

In this study, researchers will recruit 234 individuals who report binge use of alcohol or who consume alcohol moderately with no episodes of binge drinking. All participants will be recruited from the community primarily through advertisements in local newspapers, online venues like craigslist, flyers, and list-serve emails, as well as through radio and other media advertisements.

Inclusion Criteria

All Participants:

* Male and Females between the ages of 21-25
* able to read and write in English and complete study evaluations
* able to provide negative breathalyzer and negative toxicology screenings for substances at all study appointments
* able to provide written and verbal consent.
* Must be a beer drinker (not exclusively), to ensure subjects are not averse to the taste of beverages presented in the ATT
* BMI of 18-35

Binge Drinkers:

• At least twice per month binge drinking and weekly alcohol use of at least 8 standard drinks/week females or 15 or more drinks for males for the past year, with binge drinking defined as drinking enough alcohol that brings blood alcohol concentration to 0.08 percent or higher in about 2 hours, which is typically equivalent to consuming 5 or more drinks for males, or 4 or more drinks for females.

Social Drinkers:

• at least weekly alcohol use for the past 6 months not to exceed 7 standard drinks/wk for women and 14 standard drinks/week for males, with no episodes of binge drinking in the past year

Exclusion Criteria:

All Participants:

* Any psychotic disorder or current psychiatric symptoms requiring specific attention, including active symptoms of psychosis or suicidal/homicidal ideation
* meets criteria for current or past moderate or severe substance use disorder
* women who are pregnant or lactating
* inability to give informed consent
* any contraindications for MRI (e.g., medical devices in the body, claustrophobia, etc)
* current PTSD or acute stress disorder
* other illicit drug use as determined by a urine drug screen

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 234 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Neural cue reactivity to alcohol stimuli (fMRI BOLD response) | Baseline, 1-year follow-up, 2-year follow-up.
  Change in blood-oxygen-level dependent (BOLD) activation to alcohol versus neutral cues in regions of interest (e.g., medial prefrontal cortex, posterior cingulate cortex, striatum) measured using 7 Tesla functional MRI.
Cortisol and IL-6 reactivity to alcohol cues | Baseline, 1-year follow-up, 2-year follow-up.
  Change in plasma cortisol and interleukin-6 concentrations (pg/mL) from pre- to post-cue exposure in the laboratory alcohol administration session.
Alcohol craving and consumption following cue exposure | Baseline, 1-year follow-up, 2-year follow-up.
  Alcohol craving ratings on the Alcohol Urge Questionnaire (1-7 visual analog scale, high scores mean worse outocme) and total volume of alcohol consumed (mL) during the Alcohol Taste Test following cue exposure.

SECONDARY OUTCOMES:
Real-world craving and drinking behavior (EMA) | 30-day EMA period after each assessment wave (baseline, 1 year, 2 years).
  Ecological Momentary Assessment (EMA) measures of craving, alcohol use, and contextual factors collected via smartphone app 3-5 times daily for 30 days following each lab session.
Composite biomarker index of neurobiological vulnerability | Baseline, 1-year follow-up, 2-year follow-up.
  Composite score derived from standardized z-scores across neural, neuroendocrine, and immune cue-reactivity measures representing multi-attribute vulnerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University MRI Center, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will generate de-identified multimodal data from 234 participants (sex-balanced binge and non-binge alcohol users), including demographics, questionnaires, EMA (stress, craving, drinking), fMRI alcohol cue-reactivity data, cortisol and IL-6 assays, and Alcohol Taste Test results. De-identified participant-level data, survey instruments, codebooks, and metadata (DDI-compliant PDFs) will be shared via the NIDA-funded ICPSR-NAHDAP repository. MRI data will be defaced and formatted in BIDS; other data will be in .csv format, processed using R, FSL, Freesurfer, Matlab, SAS, SPSS, and Mplus, following ICPSR documentation standards. Data will be deposited within two years of project completion (or publication) and maintained in perpetuity. Access will be restricted to qualified researchers under a data-use agreement and IRB approval, with all identifiers stored separately. The PI will oversee compliance and privacy protections under NIH Certificate of Confidentiality.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available in 2033 and remain accessible thereafter.